CLINICAL TRIAL: NCT00998270
Title: A Prospective, Randomized Trial of Autologous Bone Marrow Transplantation Compare With Allogeneic Bone Marrow Transplantation in Multiple Myeloma
Brief Title: Autologous Bone Marrow Transplantation (BMT) Compared With Allogeneic BMT in Multiple Myeloma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HORCSCT-0901
Record Dates: First submitted 2009-10-17; First posted 2009-10-20 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma
Keywords: MM
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous arm (Active Comparator)
  Interventions: Procedure: Autologous bone marrow transplantation
- Allogeneic arm (Experimental)
  Interventions: Procedure: Allogeneic bone marrow transplantation

INTERVENTIONS:
Procedure: Autologous bone marrow transplantation — Autologous transplantation:
  * Endoxan (for mobilization) Dose: 2.5 g/m2 IV Time: -11 Duration: 1 day
  * G-CSF (Neupogen) Dose: 0.5 micg/kg subcutaneous Time: -6 to -3 Duration: 4 days
  * Melphalan Dose: 100 mg/m2 IV Time: -2 and -1 Duration: 2 days
  Other Names: Autologous
  Arms: Autologous arm
Procedure: Allogeneic bone marrow transplantation — Allogeneic
  * Melphalan Dose: 70 mg/m2 IV Time: Duration: 2 days
  * Fludarabine Dose: 30 mg/m2 IV Time: Duration: 5 days
  Other Names: Allogeneic
  Arms: Allogeneic arm

SUMMARY:
A prospective, randomized trial of autologous bone marrow transplantation compared with allogeneic bone marrow transplantation in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis equal or under 55 year
* Meeting the Durie and Salmon criteria for initial diagnosis of MM
* Stage II or III MM at diagnosis or anytime thereafter
* Symptomatic MM requiring treatment at diagnosis or anytime thereafter
* If receiving chemotherapy-based mobilization regimens, must be able to receive high-dose melphalan between 2 and 8 weeks after the initiation of mobilization therapy whether delivered at the transplant center or at a referring center
* Adequate organ function as measured by:

  * Cardiac: Left ventricular ejection fraction at rest greater than 40%
  * Hepatic: Bilirubin less than 2 times the upper limit of normal and ALT and AST less than 3 times the upper limit of normal
  * Renal: Creatinine clearance greater than 40 ml/min (measured or calculated/estimated)
  * Pulmonary: DLCO, FEV1, and FVC greater than 50% of predicted value (corrected for hemoglobin), or O2 saturation greater than 92% of room air
* An adequate autologous graft defined as a cryopreserved PBSC graft containing at least 4.0 x 10^6 CD34+ cells/kg patient weight; if prior to enrollment it is known that a patient will be on the auto-allo arm (i.e., a consenting, eligible HLA-matched sibling donor is available), the required autograft must contain at least 2.0 x 10^6 CD34+ cells/kg patient weight; the graft may not be CD34+ selected or otherwise manipulated to remove tumor or other cells; the graft can be collected at the transplanting institution or by a referring center; for patients without an HLA-matched sibling donor, the autograft must be stored so that there are two products each containing at least 2 x 10^6 CD34+ cells/kg patient weight

Exclusion Criteria:

* Never advanced beyond Stage I MM since diagnosis
* Non-secretory MM (absence of a monoclonal protein [M protein] in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques)
* Plasma cell leukemia
* Karnofsky performance score less than 70%, unless approved by the Medical Monitor or one of the Protocol Chairs
* Uncontrolled hypertension
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms)
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Medical Monitor or one of the Protocol Chairs; cancer treated with curative intent more than 5 years previously will be allowed
* Pregnant or breastfeeding
* Seropositive for the human immunodeficiency virus (HIV)
* Unwilling to use contraceptive techniques during and for 12 months following treatment
* Prior allograft or prior autograft
* Received mid-intensity melphalan (more than 50 mg IV) as part of prior therapy
* Prior organ transplant requiring immunosuppressive therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival and Progressive Free Survival in both two arms | 1 year

SECONDARY OUTCOMES:
Overall Survival and Progressive Free Survival in both two arms | 3 year
Treatment Related Mortality (TRM) in both two arms | 3 year
Acute and Chronic GVHD in Allogeneic arm | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Ghavamzadeh, MD, Principal Investigator — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran